CLINICAL TRIAL: NCT05912517
Title: A Phase 3 Randomized, Placebo-Controlled, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of Nipocalimab in Pregnancies at Risk for Severe Hemolytic Disease of the Fetus and Newborn (HDFN)
Brief Title: A Study of Nipocalimab in Pregnancies at Risk for Severe Hemolytic Disease of the Fetus and Newborn (HDFN)
Acronym: AZALEA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR109199; 80202135EBF3001 (Other: Janssen Research & Development, LLC); 2021-002359-12 (EudraCT Number); 2022-502629-16-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hemolytic Disease of the Fetus and Newborn

STUDY DESIGN:
Intervention Model Description: The participants will be randomized in a 2:1 to receive nipocalimab and placebo treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nipocalimab (Experimental): Participants will receive nipocalimab intravenously (IV) once weekly (qw) from randomization through gestational age (GA) Week 35.
  Interventions: Drug: Nipocalimab
- Placebo (Placebo Comparator): Participants will receive matching placebo IV qw from randomization through GA Week 35.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nipocalimab — Nipocalimab will be administered as an intravenous infusion.
  Other Names: JNJ-80202135; M281; JNJ-86507083
  Arms: Nipocalimab
Drug: Placebo — Placebo will be administered as an intravenous infusion.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness of nipocalimab when compared to placebo in decreasing the risk of fetal anemia (a condition in which a baby's red blood cell volume falls below normal levels while the baby is developing in the womb) with live neonates in pregnant participants at risk for severe hemolytic disease of the fetus and newborn.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and an estimated gestational age (GA) (based on ultrasound dating) from Week 13^0/7 to Week 18^6/7 at randomization
* History of severe Hemolytic Disease of the Fetus and Newborn (HDFN) in a prior pregnancy defined as documented:

  1. fetal anemia as result of HDFN or fetal hydrops as result of HDFN or received greater than or equal to (>=)1 IUT as a result of HDFN or
  2. fetal loss or neonatal death as a result of HDFN, with maternal alloantibody titers for Rhesus antigen D protein (RhD), Kell, Kell Rhesus antigen C protein (Rhc), Rhesus antigen E protein (RhE), or RhC antigen above the critical levels (anti-Kell >=4; other >=16) and evidence of an antigen-positive fetus
* During the current pregnancy, presence of maternal alloantibody to RhD, Rhc, RhE, or RhC antigen with titers above the critical level (anti-Kell >= 4; other >=16) based on the designated central lab results at screening
* Evidence of antigen-positivity corresponding to the current maternal alloantibody (RhD, Kell, Rhc, RhE, or RhC) confirmed by non-invasive antigen cell-free fetal DNA (cffDNA) performed at the central laboratory
* Have screening lab test results within values within the study protocol-specified parameters: a) albumin >= lower limit of normal (LLN); b) alanine transaminase (AST) less than or equal to (<=) 2 × upper limit of normal (ULN); c) alanine transaminase (ALT) <=2 × ULN d) creatinine <=0.8 milligrams per deciliter (mg/dL), SI: <=70.7 micromole per liter (μmol/L), and Serum total immunoglobulins G (IgG) ≥ 600 mg/dL SI: >=6 g/L
* Medically stable on the basis of physical examination, medical history, vital signs, 12-lead ECG, and clinical lab tests performed at screening

Exclusion Criteria:

* Currently pregnant with a multiple gestation (twins or more)
* Evidence of fetal anemia prior to randomization in the current pregnancy
* History of severe preeclampsia prior to GA Week 34 or severe fetal growth restriction (estimated fetal weight <3rd percentile, based on local fetal growth normative standards) in a previous pregnancy
* Current uncontrolled hypertension
* History of myocardial infarction, unstable ischemic heart disease, or stroke
* Has any confirmed or suspected clinical immunodeficiency syndrome or has a family history of congenital or hereditary immunodeficiency unless confirmed absent in the participant
* Has inflammatory or autoimmune diseases requiring immunosuppressive therapies that may jeopardize the safety of the participant
* Currently has a malignancy or has a history of malignancy within 3 years before screening (with the exception of localized basal cell carcinoma and/or squamous cell carcinoma skin cancer that has been adequately treated with no evidence of recurrence for at least 3 months before the first study intervention administration or cervical carcinoma in situ that has been treated with no evidence of recurrence for at least 3 months before the first study intervention)
* Is currently receiving systemic corticosteroids or other immunosuppressants for disorders unrelated to the pregnancy
* Has received or planning to receive plasmapheresis, immunoadsorption therapy, intravenous immunoglobulin (IV Ig), or any immunoglobulin (Ig)G fragment crystallizable (Fc)-related protein therapeutics during the current pregnancy
* Has a severe infection including opportunistic infections
* Presence of abnormal (protocol-specified) hematologic lab values during screening
* History of an unprovoked pulmonary embolism or history of recurrent deep vein thrombosis (DVT)

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2027-08-05 (Estimated); Study Completion 2029-07-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Pregnancies That did not Result in Fetal Loss, Intrauterine Transfusion (IUT), Hydrops Fetalis, or Neonatal Death | From randomization in the study through 4 weeks of age or 41 weeks Postmenstrual Age (PMA) during neonatal period, whichever is later
  Percentage of pregnancies that did not result in fetal loss, IUT, hydrops fetalis, or neonatal death (during the neonatal period) will be reported. Hydrops fetalis is defined as the presence of greater than or equal to(>=)2 abnormal fluid collections in the fetus or neonate, such as ascites, pleural effusions, pericardial effusion, and generalized skin edema (skin thickness greater (>)5 millimeter [mm]). PMA is the time elapsed between the first day of the last menstrual period and birth (gestational age) plus the time elapsed after birth (chronological age).

SECONDARY OUTCOMES:
Number of Participants With Hemolytic Disease of the Fetus and Newborn (HDFN) by Severity | For first database lock: from randomization in the study through 4 weeks of age or 41 weeks PMA during neonatal period, whichever is later for the first database lock; for second database lock: through 12 weeks after birth
  Number of participants with HDFN by severity will be reported. The severity of HDFN is defined as: 5 (fatal): fetal or neonatal death due to any reason; 4 (severe): hydrops fetalis (in fetus or newborn) or receiving IUT during pregnancy as a result of HDFN but not 5 (fatal); 3 (moderate): neonatal exchange transfusions received as a result of HDFN related hemolysis and jaundice but not 4 (severe) or 5 (fatal); 2 (mild): neonatal simple transfusions received due to HDFN after birth, with or without phototherapy, but not 3 (moderate), 4 (severe), or 5 (fatal); and 1 (minimal or none): not in 2 (mild), 3 (moderate), 4 (severe), or 5 (fatal) as described above. Here database lock implies the last participant has given birth or terminated their pregnancy, completed the Week 4 visit after delivery, and whose neonate has also completed the Week 4 visit (or 41 weeks PMA, whichever is later) or died prior to this timepoint.
Time to First Occurrence of IUT or Hydrops Fetalis | From randomization to delivery of baby (Up to 38 weeks)
  Time to first occurrence of IUT or hydrops fetalis will be reported.
Neonatal Mortality and Morbidity Index (NMMI) in Liveborn Neonates | Through 38 weeks PMA or at discharge if earlier than 38 weeks PMA
  The NMMI will be assessed with the following categories: fatal: fetal/neonatal death; major morbidity: any of intraventricular hemorrhage grade 3/4, seizures, hypoxic-ischemic encephalopathy, necrotizing enterocolitis stage 2/3, respiratory distress syndrome requiring mechanical ventilation, bronchopulmonary dysplasia requiring oxygen support, or persistent pulmonary hypertension; Minor morbidity: anemia requiring simple transfusion, hyperbilirubinemia requiring an exchange transfusion, hypotension requiring treatment, intraventricular hemorrhage grade 1/2, necrotizing enterocolitis stage 1, or respiratory distress syndrome not requiring mechanical ventilation; None: no major or minor morbidities described above. Hyperbilirubinemia requiring phototherapy will be classified in this category'
Number of IUT's Received During the Pregnancy | From randomization to delivery of baby (Up to 38 weeks)
  Number of IUT's received during the pregnancy will be reported.
Percentage of Pregnancies With Fetal Loss | Time to delivery of baby (Up to 38 weeks)
  Percentage of pregnancies with fetal loss will be reported.
Percentage of Pregnancies With Fetal or Neonatal Death | Through Week 4 or 41 weeks PMA
  Percentage of pregnancies with fetal or neonatal death (through the neonatal period) as a result of HDFN will be reported.
Percentage of Pregnancies With Hydrops Fetalis | Up to 41 weeks PMA
  Percentage of pregnancies with hydrops fetalis will be reported. Hydrops fetalis is defined as the presence of >=2 abnormal fluid collections in the fetus or neonate, such as ascites, pleural effusions, pericardial effusion, and generalized skin edema (skin thickness >5 mm).
Percentage of Pregnancies Receiving IUT During Pregnancy | Up to 35 weeks of GA period
  Percentage of pregnancies receiving IUT during pregnancy will be reported.
Gestational Age (GA) at First IUT | Up to 35 weeks of GA period
  GA at first IUT will be reported.
Percentage of Pregnancies Receiving >1 IUT During Pregnancy | Up to 35 weeks of GA period
  Percentage of pregnancies receiving >1 IUT during pregnancy will be reported.
Percentage of Pregnancies Receiving IUT or HDFN Resulting in Fetal Demise (Less Than) <GA Week 20 | Up to 20 weeks
  Percentage of pregnancies receiving IUT or HDFN resulting in fetal demise <GA Week 20 will be reported.
Gestational Age at Delivery | Up to 38 weeks
  Gestational age at delivery will be reported.
Percentage of Pregnancies With Neonatal Death Through the Neonatal Period | From randomization in the study through 4 weeks of age or 41 weeks PMA during neonatal period, whichever is later
  Percentage of pregnancies with neonatal death through the neonatal period will be reported.
Percentage of Liveborn Neonates With HDFN-related Morbidities Other Than Anemia and Hyperbilirubinemia or Jaundice | From day of birth up to 4 weeks
  Percentage of liveborn neonates with HDFN-related morbidities other than anemia and hyperbilirubinemia or jaundice will be reported.
Absolute Weight of Liveborn Neonates or Infants | Up to 104 weeks
  Absolute weight of liveborn neonates or infants will be reported.
Change From Baseline in Weight of Liveborn Neonates or Infants | Baseline to up to 104 weeks
  Change from baseline in weight of liveborn neonates or infants will be reported.
Liveborn Neonates Length of Stay in Neonatal Intensive Care Unit | From day of birth up to 27 days
  Liveborn neonates length of stay in neonatal intensive care unit will be reported.
Percentage of Liveborn Neonates Receiving Exchange Transfusions for HDFN | From day of birth up to 27 days
  Percentage of liveborn neonates receiving exchange transfusions for HDFN will be reported.
Number of Neonatal Exchange Transfusions per Liveborn Neonate | From day of birth up to 27 days
  Number of neonatal exchange transfusions per liveborn neonate will be reported.
Percentage of Liveborn Neonates or Infants with Simple Transfusions for HDFN | For first database lock: From birth up to 4 weeks; for second database lock: From birth up to 12 weeks
  Percentage of liveborn neonates or infants with simple transfusions for HDFN through the neonatal period (for the first database lock) or 12 weeks (for the second database lock) after birth will be reported.
Number of Simple Transfusions for HDFN per Liveborn Neonate or Infant | For first database lock: From birth up to 4 weeks; for second database lock: From birth up to 12 weeks
  Number of simple transfusions for HDFN per liveborn neonate or infant through the neonatal period (for the first database lock) or 12 weeks (for the second database lock) after birth will be reported.
Percentage of Liveborn Neonates With Hyperbilirubinemia Treated With Phototherapy | From day of birth up to 27 days
  Percentage of liveborn neonates with hyperbilirubinemia treated with phototherapy will be reported.
Number of Days of Phototherapy Received for Hyperbilirubinemia per Liveborn Neonate | From day of birth up to 27 days
  Number of days of phototherapy received for hyperbilirubinemia per liveborn neonate will be reported.
Percentage of Liveborn Neonates or Infants Receiving Intravenous Immunoglobulin (IVIg) for HDFN Treatment | For first database lock: From birth up to 4 weeks; for second database lock: From birth up to 12 weeks
  Percentage of liveborn neonates or infants receiving IVIg for HDFN treatment will be reported.
Number of Maternal Deaths | Form randomization up to 24 weeks postpartum
  Number of maternal deaths will be reported.
Number of Participants with Adverse Events (AEs) | From randomization up to 24 weeks postpartum
  Number of participants with AEs, serious adverse events, and AEs of special interest (AESIs), AE's leading to discontinuations, infections, serious infections, infusion reactions, and hypersensitivity reactions will be reported. Treatment-emergent adverse events associated with the following situations are considered as AESIs: hypoalbuminemia, clinically significant bleeding with a corresponding placental finding on ultrasound, maternal infections that led to clinically significant morbidities or mortalities in fetus or neonates, Infections that are severe or require intravenous (IV) anti-infective or operative or invasive intervention in maternal participants or neonates or infants, and infants with hypogammaglobulinemia.
Number of Maternal Pregnancy Complications | Up to 38 weeks
  Number of maternal pregnancy complications will be reported.
Number of IUT Related complications | Up to 35 weeks of GA period
  Number of participants with IUT related complications will be reported.
Percentage of Pregnancies With Cesarean Delivery, Preterm Birth, Fetal Growth, and Preeclampsia | Up to 38 weeks of GA period
  Percentage of pregnancies with cesarean delivery, cesarean delivery due to IUT complications, preterm birth <GA week 28, preterm birth <GA week 32, preterm birth <GA week 34, preterm birth <GA week 37, fetal growth restriction, and preeclampsia will be reported.
Percentage of Liveborn Neonates or Infants Who Died | Up to 104 weeks
  Percentage of liveborn neonates or infants who died will be reported.
Percentage of Liveborn Neonates or Infants With AEs | Up to 104 weeks
  Percentage of liveborn neonates or infants with AEs, SAEs, AESIs, infections, serious infections will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. Any event requiring hospitalization (or prolongation of hospitalization) that occurs during participation in the study must be reported as an SAE.
Percentage of Liveborn Neonates or Infants Receiving IVIg for Non-HDFN Indications | Up to 104 weeks
  Percentage of liveborn neonates or infants receiving IVIg for non-HDFN indications will be reported.
Percentage of Liveborn Neonates or Infants With Abnormal Hearing | Up to 104 weeks
  Percentage of liveborn neonates or infants with abnormal hearing will be reported.
Bayley Scales of Infant Development and Toddler Development | Week 52 and 104
  The Bayley Scales of infant development is considered the standard assessment of early child development and includes cognition, language, motor skills, social emotional, and adaptive behavior will be reported. The Bayley Scales (3rd edition) are reference standards that measure infant and toddler development in five areas: cognition, language, motor skills, social-emotional and adaptive behavior. The cognition, language and motor skills scales are directly administered to the infant, while social-emotional, and adaptive behavior scales are caregiver questionnaires. The scores are standardized using norm reference samples with representative demographics and age adjusted for prematurity. Higher scores in the Bayley Scales indicate better outcomes.
Change From Baseline in Generalized Anxiety Disorder 7-Item (GAD7) Over time During Pregnancy and Postpartum | Baseline (Day 1) and Week 30 during pregnancy and Week 4 postpartum
  Change from baseline in GAD7 over time during pregnancy and postpartum will be reported. The GAD-7 scale is a self-administered questionnaire designed to measure anxiety. The recall period for all items is the past 2 weeks. Responses to all items are rated on a 4-point Likert scale ranging from 0 "not at all" to 3 "nearly every day". The total score ranges from 0 to 21, with higher scores indicating higher severity of anxiety symptoms.
Change From Baseline in Short Form 36 Version 2 (SF-36v2) Acute Form Domain Score | Baseline (Day 1) and Week 30 during pregnancy and Week 4 postpartum
  Change from baseline in SF-36v2 acute form domain score will be reported. The SF-36 version 2 acute is a self-administered, 36-item questionnaire measuring health-related quality of life and includes 8 domains that measure physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality social functioning, role limitations due to emotional problems, and mental health. The 8 domains can be aggregated into 2 summary scales that reflect physical and mental health: a physical component summary and a mental component summary. Responses to all items are rated on a 3, 5, or 6-point Likert scale, with higher scores indicating better health status.
Change From Baseline in EuroQol Five-dimension Questionnaire (EQ-5D-5L) Visual Analogue Scale (VAS) Score | Baseline (Day 1) and Week 30 during pregnancy and Week 4 postpartum
  Change from baseline in EQ-5D-5L visual analogue score will be reported. The EQ-5D descriptive system is comprised of 5 items across the following 5 dimensions: mobility, self-care, usual activities, pain or discomfort and anxiety or depression. The EQ-5D-5L uses a 5-point Likert response scale ranging from "no problems" to "extreme problems", with higher scores indicating better quality of life. EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ-VAS). EQ-VAS score ranges from 0 to 100, where 0 = worst imaginable health state and 100 = best imaginable health state. Higher score indicates good health state.
Change From Baseline in EuroQol 5-Dimension Descriptive (EQ-5D) Index Score | Baseline (Day 1) and Week 30 during pregnancy and Week 4 postpartum
  Change from baseline in EQ-5D index score will be reported. The EQ-5D descriptive system is comprised of 5 items across the following 5 dimensions: mobility, self-care, usual activities, pain or discomfort and anxiety or depression. The EQ-5D-5L descriptive system uses a 5-point Likert response scale ranging from "no problems" to "extreme problems", with higher scores indicating better quality of life.
Infant Health-Related Quality of Life Instrument (IQI) Score for Neonate or Infant Overtime | Weeks 4, 8 and 52
  IQI score for neonate or infant will be reported. The IQI consists of 7 health attributes including sleeping, feeding, breathing, stooling or poo, mood, skin, and interaction. Responses to all items are rated on a 4-point Likert scale, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (57):
- United States (16):
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - UC Davis School of Medicine, Sacramento, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Advocate Children's Hospital, Park Ridge, Illinois
  - Riley Children s Hospital, Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Midwest Fetal Care Center, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - University of North Carolina (UNC) - School of Medicine, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - University of Texas Dell Medical School Department of Women's Health, Austin, Texas
  - University Of Texas Medical Branch At Galveston, Galveston, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
- Argentina (2):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Privado Universitario De Cordoba, Córdoba
- Australia (2):
  - Mater Hospital Brisbane, South Brisbane
  - Liverpool Hospital, Sydney
- Medizinische Universitaet Wien, Vienna, Austria
- Belgium (2):
  - C.H.U. Brugmann, Brussels
  - Universitair Ziekenhuis Leuven, Leuven
- Brazil (5):
  - Universidade Federal De Minas Gerais, Belo Horizonte
  - Empresa Brasileira de Servicos Hospitalares EBSERH Hospital das Clinicas da UFG, Goiânia
  - Instituto de Medicina Integral Professor Fernando Figueira, Recife
  - Instituto D Or de Pesquisa e Ensino IDOR, Rio de Janeiro
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Canada (3):
  - BC Women's Hospital University of British Columbia, Vancouver, British Columbia
  - Centre Hospitalier Sainte Justine, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- France (3):
  - Hospices Civils de Lyon - Groupement Hospitalier Est - Hopital Femme Mere Enfant, Bron
  - CHRU Lille, Lille
  - Hopital Armand Trousseau, Paris
- Germany (2):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Giessen und Marburg Standort Giessen, Giessen
- Rotunda Hospital, Dublin, Ireland
- Israel (3):
  - Hadassah mount scopus, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
- Fondazione Policlinico Universitario A Gemelli IRCCS, Roma, Italy
- Japan (5):
  - Kyushu University Hospital, Fukuoka
  - Gifu Prefectural General Medical Center, Gifu
  - Osaka Women's and Children's Hospital, Izumi-shi
  - Toho University Medical Center Omori Hospital, Ōta-ku
  - Miyagi Children's Hospital, Sendai
- Leiden University Medical Center, Leiden, Netherlands
- Spain (3):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Virgen Del Rocio, Seville
- Karolinska Universitetssjukhuset Huddinge, Stockholm, Sweden
- United Kingdom (6):
  - Birmingham Women's Hospital, Birmingham
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Kings College Hospital, London
  - St Georges Hospital, London
  - St.Mary's Hospital, Manchester
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Rego S, Ashimi Balogun O, Emanuel K, Overcash R, Gonzalez JM, Denomme GA, Hoskovec J, King H, Wilson A, Wynn J, Moise KJ Jr. Cell-Free DNA Analysis for the Determination of Fetal Red Blood Cell Antigen Genotype in Individuals With Alloimmunized Pregnancies. Obstet Gynecol. 2024 Oct 1;144(4):436-443. doi: 10.1097/AOG.0000000000005692. Epub 2024 Jul 25. PMID 39053010
- See also: Azalea Study Website (for the United States only) — https://azaleatrial.com
- See also: Participant Recruitment Poster — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR109199&attachmentIdentifier=cb7c7ecc-ba54-4995-bc49-030c76585fcc&fileName=80202135EBF3001_ENG20_Participant_Recruitment_Poster_V1.0_9Mar2023.pdf&versionIdentifier=